CLINICAL TRIAL: NCT04516954
Title: Assessment of the Safety of Convalescent Plasma to Treat COVID-19 Patients With Moderate and Above Illness
Brief Title: Convalescent Plasma for COVID-19 Patients
Acronym: CPCP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Collaborators: National Institute of Hygiene and Epidemiology, Vietnam (Other); National Hospital for Tropical Diseases, Hanoi, Vietnam (Other Government); National Institute of Hematology and Blood Transfusion, Vietnam (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISC.20.11.1
Record Dates: First submitted 2020-08-17; First posted 2020-08-18 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Convalescent COVID 19 Plasma (Experimental): A total of 500 ml of convalescent COVID 19 plasma will be transfused intravenously per subject
  Interventions: Biological: Convalescent COVID 19 Plasma

INTERVENTIONS:
Biological: Convalescent COVID 19 Plasma — A total of 500 ml of convalescent COVID 19 plasma will be transfused intravenously per subject

SUMMARY:
The investigators propose to evaluate intravenous administration of convalescent plasma (CP) obtained from COVID19 survivors in COVID19 patients who are in the medium stage. Supportive data exist for use of convalescent plasma in the treatment of COVID19 and other overwhelming viral illnesses. The study team wants to test the hypothesis that treatment with COVID19 CP will demonstrate salutary effects on COVID19 disease severity/duration, with the primary objective to reduce mortality. In addition, a major secondary objective to reduce the requirement for and/or duration of mechanical ventilation. The first phase is to test the safety of CP therapy.

DETAILED DESCRIPTION:
Coronaviruses are among the most common causes of the common cold in humans.1,2 In recent decades, coronavirus has caused several epidemic worldwide with a vast number of deaths such as severe acute respiratory syndrome-SARS (2003) with 8098 people infected and 774 people died over 29 countries. The disease caused by SARS CoV-2 (COVID19) is manifest by fever, fatigue, dry cough, pharyngitis, and headache. In addition to the common clinical presentation of respiratory distress, and increasing frequency of cardiovascular manifestations has become evident.

In this context, the investigators propose to evaluate the safety of intravenous administration of convalescent plasma (CP) obtained from COVID19 survivors in patients requiring hospitalization for symptomatic "high risk" COVID19 disease. The study team wants to test the hypothesis that treatment with COVID19 CP will demonstrate salutary effects on COVID19 disease severity/duration, with the primary objective to reduce mortality. In addition, a major secondary objective to reduce the requirement for and/or duration of mechanical ventilation This is a single-arm, non-randomized, open-label treatment of eligible subjects defined as those who satisfy all inclusion criteria.

Written informed consent will be obtained all eligible subjects prior to participation.

Convalescent plasma will be obtained from male donors, nulliparous females, or female donors negative for HLA antibodies at least 14 days following recovery from COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* SARS-CoV-19 PCR positive
* Medium stage
* Time from onset to screening ≤ 21 days, the SARS-CoV-2 test is still positive

Exclusion Criteria:

* Patients with a history of autoimmune disease or IgA deficiency
* Patients with a history of allergy
* Multi-organ/system failure
* Pregnant or breastfeeding at the time of study
* Cancer, history of heart failure, stroke, bronchial asthma
* Multi-organ/system failure with indications for dialysis, severe hypoxia, failure with conventional treatment methods, indications for ECMO.
* The patient is infected with multidrug-resistant bacteria.
* The patient is participating in another study.
* Time from onset to screening> 21 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety | At Day 28
  Number of Adverse Events (AEs), and Serious Adverse Events (SAEs) of COVID 19 Patients:
  Incidence of Treatment-Emergent Adverse Events (Data on the number of participants with treatment related adverse events will be assessed to determine the safety and tolerability of convalescent plasma)

SECONDARY OUTCOMES:
Change in requirement for mechanical ventilatory support | At Day 28
  Change in the duration of mechanical ventilation in COVID 19 patients compared with historic precedent cohorts

CONTACTS AND LOCATIONS:
Locations (1):
- Vinmec Research Institute of Stem cell and Gene Technology, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No